CLINICAL TRIAL: NCT02591459
Title: Android Mobile Devices to Assist Routine Anticipation for Autistic Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Annie France Frère Slaets, PhD, University of Mogi das Cruzes
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 49354415.0.0000.5497
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Autism
Keywords: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autism (Other): Using the app to assist routine anticipation for autistic children in Android mobile devices
  Interventions: Other: Using the app to assist routine anticipation

INTERVENTIONS:
Other: Using the app to assist routine anticipation — Using the app to assist routine anticipation for autistic children in Android mobile devices

SUMMARY:
The objective of this work is to develop an application to run on a mobile device Android tablet that features visual routines for autistic children.

DETAILED DESCRIPTION:
Autism is a disorder characterized by social deficits, and among others by changes in communication. The diagnosis of this disorder remains accomplished by direct assessment the individual's behavior, according to specific clinical criteria present the classification systems of the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV). Therapists teach autistic to communicate with the help of symbols and auxiliary anticipation and communication routines, usually using the Picture Exchange Communication System (PECS), or photos. However these are presented in transition PECS cards and do not follow the children in activities that develop outside the school environment. The objective of this work is to develop an application to run on a mobile device Android tablet that features the visual routines.

In this way the routines can be accessed outside the school environment. This technology is easy to use and facilitates data entry by touching the screen, was developed using the Unified Modeling Language (UML), Javascript, Apache Web server and Web browser Chrome. The application validation, will be held with 10 autistic and 2 teachers from the center of inclusion and support for autistic. Teachers should insert the activities programmed for each autistic student. Tablet in student performance in communicating with this tablet will be measured. Parents or guardians knowledge with the PECS system will be trained and will be evaluated on their autonomy inserting images, audio and subtitles. The application should aid communication, cause the autistic understand the sequence of events in daily life, decreasing their aggression because of not knowing what will be their next activity. Participation in this research poses no risk or harm the concerned person. If during the research participant decides not anymore have the freedom to do so without incurring any damage you. The technical validation proposal is necessary for it to be used by people with autism. If validated in a positive way, the technique could improve the quality of life of these people and their families.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of autism development by DSM-IV
* Have sufficient motor skills to perform operations on a tablet
* Be aware of PECS
* Children should be accustomed to the visual routines used in

Exclusion Criteria:

* Have visual impairment

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Increase in verbal communication | 1 month
  Increased verbal communication in autistic individuals (as a percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Annie F Frere Slaets, PhD, Principal Investigator — University of Mogi Cruzes
Locations (1):
- Centro de inclusão e Apoio ao Autista de Guarulhos (CIAAG), Guarulhos, São Paulo, Brazil